CLINICAL TRIAL: NCT01327690
Title: Mental Health in Veterans and Families After Group Therapies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Principal Investigator, Dawson Church, Principal Investigator, Soul Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: SMI-GROUP-12/10/10
Record Dates: First submitted 2011-01-04; First posted 2011-04-01 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Post-Traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Wait List (No Intervention): Wait Period corresponding in length to treatment period
- EFT (Emotional Freedom Techniques) (Experimental): EFT group therapy sessions.
  Interventions: Behavioral: EFT (Emotional Freedom Techniques)
- CBT (Cognitive Behavior Therapy) (Active Comparator): CBT group therapy sessions
  Interventions: Behavioral: CBT (Cognitive Behavior Therapy)

INTERVENTIONS:
Behavioral: CBT (Cognitive Behavior Therapy) — CBT group therapy sessions
  Arms: CBT (Cognitive Behavior Therapy)
Behavioral: EFT (Emotional Freedom Techniques) — Group therapy sessions using EFT
  Arms: EFT (Emotional Freedom Techniques)

SUMMARY:
PTSD (posttraumatic stress disorder) and associated mental health conditions affect both veterans and their family members. This study investigates whether group therapy using EFT (Emotional Freedom Techniques) and CBT (Cognitive Behavior Therapy) produce reductions in PTSD and comorbid symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The ability to follow instructions, complete written forms, and provide informed consent. Subjects are required to be literate and understand English.
* Physically healthy.
* Active duty military service, veterans, and their family members.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline PTSD (posttraumatic stress disorder) Symptom Levels | Pre-Intervention, Post-Intervention, with one, three, six, and twelve month follow-ups
  Symptoms are measured before the first group therapy session. Symptom levels are also recorded immediately after the last group session, and at follow-up points: one, three, six, and twelve months later.

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Principal Investigator — Soul Medicine Institute
Locations (1):
- Soul Medicine Institute, Santa Rosa, California, United States

REFERENCES:
- See also: Related Info — http://www.NIIH.org/